CLINICAL TRIAL: NCT04941001
Title: Optimisation of ASthma In Those With Uncontrolled Symptoms (OASIS) in Primary Care Using a Digital Consultation Tool During the COVID-19 Pandemic
Brief Title: Optimisation of ASthma In Those With Uncontrolled Symptoms (OASIS)
Acronym: OASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 274450
Record Dates: First submitted 2021-06-03; First posted 2021-06-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-07

CONDITIONS: Asthma; Asthma Attack; Asthma Persistent; Covid19
MeSH Terms: conditions — Asthma; COVID-19

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: An electronic randomisation programme will be used to assign the patient to each arm of the study in primary care. However during the review, masking will not be possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthcare professional using ReferID Tool in primary care (Active Comparator): The asthma review will be undertaken by a healthcare professional with the use of the ReferID tool in primary care
  Interventions: Device: ReferID
- Usual care in primary care (No Intervention): A cohort of patients will be recruited who continue to receive usual care in primary care

INTERVENTIONS:
Device: ReferID — The ReferID tool is a digital tool which can be used to facilitate a review of asthma in primary care
  Arms: Healthcare professional using ReferID Tool in primary care

SUMMARY:
A digital tool, called ReferID has been developed to facilitate the review of asthma patients. It aims to assist in the identification of patients with uncontrolled and/or severe asthma and to ensure a timely referral to secondary care where appropriate. To validate the tool, patients will be randomised to have a review with a healthcare professional using tool to facilitate the review or to continue receiving usual care. Outcome measures including exacerbation frequency and level of asthma control will be assessed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All asthma patients with 1 of more exacerbations in the last 12 months or receiving high dose inhaled corticosteroids.
* Patients able and willing to provide informed consent.
* Patients aged 18 and over.

Exclusion Criteria:

* Patients who lack capacity.
* Patients who do not have a diagnosis of asthma
* Patients who are unable to provide informed consent
* Patients under the age of 18
* Patients already under a severe asthma centre

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Rate of exacerbation frequency | 24 months
  Measured by the number of courses of oral corticosteroids measured at 12 months before and 12 months after initial consultation. Exacerbations are defined as the need for oral corticosteroids prescribed by a healthcare professional for a minimum of 3 consecutive days in the context of worsening asthma symptoms.

SECONDARY OUTCOMES:
Asthma control measured by the Asthma Control Questionnaire (ACQ) - 6. | 12 months
  Asthma control questionnaire completed on day 1 and at 12 months after initial consultation. Total score ranges from 0-6, with 0 = no impairment due to asthma, 6 = maximum impairment due to asthma.
Salbutamol use (measured by the number of inhalers issued) | 24 months
  Change in primary care salbutamol prescription refill frequency 12 months before and 12 months after initial consultation.
Emergency care utilisation | 24 months
  Frequency of emergency department and/or hospital admission due to acute asthma 12 months before and 12 months after initial consultation.
Quality of Life Score measured by the mini Asthma Quality of Life Questionnaire (mAQLQ) | 12 months
  Change in quality of life score at day 1 and at 12 months (mAQLQ). Score for each question ranges from 0-7, with 0 = totally limited, 7 = not limited at all. The score is calculated as an average for each domain, with a clinically minimum difference of 0.5.
Adherence to inhaled corticosteroids | 24 months
  Adherence to inhaled corticosteroids 12 months before and 12 months after initial consultation (measured as a percentage of the number of doses of inhaled corticosteroids issued/the expected number of doses in 12months).
Inhaler technique assessed. | 12 months
  Proportion of subjects invited to have a review and found to have suboptimal inhaler technique.
Number of patients referred to secondary care who are taking part in the study. | 12 months
  Proportion of subjects referred to secondary care for further assessment of suspected severe asthma or work-related asthma
Number of patients initiated on biologic therapy | 12 months
  Proportion of subjects referred to secondary care with confirmed severe asthma initiated on biologic therapies
Number of patients who are found to have an incorrect diagnosis. | 12 months
  Proportion of subjects in whom the diagnosis of asthma is found to be incorrect

OTHER OUTCOMES:
Review and feedback of the ReferID Tool | 12 months
  Acceptability of using the ReferID tool by completion of questionnaire, with users providing feedback using a likert scale, with 1 = poor, 5 = excellent.

CONTACTS AND LOCATIONS:
Locations (1):
- Guys and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No